CLINICAL TRIAL: NCT03162445
Title: Bone Mass Accrual in Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ann Neumeyer, Assistant Professor Neurology, Massachusetts General Hospital
Other Study IDs: 2009P002422
Record Dates: First submitted 2017-05-12; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Autism Spectrum Disorder; Bone Diseases, Developmental
Keywords: bone mineral density; Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Bone Diseases, Developmental; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Typically developing controls: Boys between ages 7 and 14 years old at study onset without medications or diseases impairing bone development
- Autism spectrum disorder: Boys between ages 7 and 14 years old at study onset without medications or diseases impairing bone development

SUMMARY:
This is a observational study to investigate the degree to which bone mineral density is impaired in boys with autism compared with typically developing controls.

DETAILED DESCRIPTION:
Studies have shown that bone cortical thickness is decreased in children with autism and other developmental disabilities. However it is not known whether bone mineral density (BMD) of these children is lower; neither is it known whether there is any correlation between BMD and the child's diet. The overall goal of this study is to improve the long term health of children and adolescents with autism spectrum disorder; more specifically the investigators aim to develop a pilot study to investigate the degree to which BMD is impaired in boys with autism and to explore specific additional risk factors. In addition, the aim is to investigate the degree to which BMD is impaired in boys with Autism Spectrum Disorder (ASD) and to explore specific contributing risk factors including nutritional analysis.

ELIGIBILITY:
Inclusion Criteria:

* Boys 8-17 years chronological age
* BMI between the 3rd and 97th percentiles
* Meets DSM-IV criteria for Autism Spectrum Disorder (ASD group)
* Scores <15 on the Social Communication Questionnaire (control group)

Exclusion Criteria:

* Use of medications directly affecting bone metabolism including estrogen/ progesterone preparations and glucocorticoids except local application of glucocorticoid
* Use of anticonvulsants which affect bone density including diphenylhydantoin, phenobarbital, topiramate carbamazepine and valproic acid and also use of lithium
* Children with diseases known to affect bone mineral density including Crohn's disease, celiac, thyroid and renal
* Children who will not tolerate lying still for 30 seconds

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescent boys, ages 8-17 years, recruited from a clinic population (ASD) or community advertisements (ASD and control) matched for age.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Bone mineral density will be assessed within one month of enrolling in the study.
  using dual energy x-ray absorptiometry (DXA) (Hologic Discovery A, Software Version: APEX 4.0.2, Bedford, MA USA) at the total hip, femoral neck, lumbar spine (L1-4), whole body and whole body less head bone mineral density.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Neumeyer, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No